CLINICAL TRIAL: NCT06483620
Title: Neuropathy and Foot Ulcer_ Specific Quality of Life Instrument (Neuro QOL) Arabic Version: Cross-cultural Adaptation, Validity, and Reliability for Patients With Type 2 Diabetes
Brief Title: Cross-cultural Adaptation and Validity of the Arabic-translated NEUROPATHY-SPECIFIC QUALITY OF LIFE Questionnaire
Status: Recruiting | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Engy Badreldin Saleh Moustafa, PhD, Principal Investigator, Cairo University
Other Study IDs: P.T.REC/012/005051
Record Dates: First submitted 2024-06-11; First posted 2024-07-03 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2024-12

CONDITIONS: Diabetic Neuropathies; Diabetic Peripheral Neuropathy
MeSH Terms: conditions — Diabetic Neuropathies

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Diabetic Neuropathy group: The study design was a cross-cultural validation of Neuro Qol the Arabic version, for patients with DFUs. Three expert panels were involved in this study to test the face and content validity of the NeuroQol Arabic version. All experts had experience of not less than 10 years or at least a master's degree in physical therapy; a major part of their work is with the Arabic population; and they were also fluent in Arabic and English.
  Ten patients per item were chosen to estimate the sample size for testing the psychometric properties of the Neuro Qol Arabic version. So 290 patients (145 male patients and 145 female patients), were chosen according to specific eligibility criteria.
  Interventions: Diagnostic Test: Neuropathy - and Foot Ulcer - Specific Quality of Life instrument (Neuro Qol)

INTERVENTIONS:
Diagnostic Test: Neuropathy - and Foot Ulcer - Specific Quality of Life instrument (Neuro Qol) — The NeuroQoL questionnaire is a valid, reliable, and self-reported questionnaire. It has 35-items with six domains namely, painful symptoms and paresthesia (items 1-7), reduction or loss of ability to feel (items 8-10), unsteadiness while walking/standing/diffuse sensory-motor symptoms (items 11-13), limitation in daily living (items 14 - 16), interpersonal problems (items 17-20), emotional distress (items 21- 27) and end with an overall assessment of quality of life or satisfaction with experiences in the above six domains [1 item in each domains, i.e. additional 6 items (items 28-33)]. The two final items (items 34-35) assess overall impact of neuropathy on QoL [5]. The scoring of the questionnaire is according to a five-point Likert scale, all the time, most of the time, some of the time, occasionally, never. Each domain has a maximum score 5 and minimum 1, where 5 means that the QoL is affected all the time because of the foot problem while 1 means never it affects their QoL

SUMMARY:
PURPOSE: This study will translate, culturally adapt, validate, and test the reliability of the Neuro Qol Arabic version to be used with diabetic patients in Arabic countries.

Background: The Neuropathy- and Foot Ulcer-Specific Quality of Life instrument is a multidimensional scale was developed to assess the QoL of diabetic patients with peripheral neuropathy. Producing Arabic versions of the Translating Scale can help researchers investigate offloading treatment among the Arabic population with DFUs.

Hypotheses: The study design was a cross-cultural validation of NeuroQol, the Arabic version, for patients with DFUs.

Research Question: Will there be cultural adaptation, validation, and reliability between the (Neuro Qol) Arabic version and the original language?

DETAILED DESCRIPTION:
The Neuropathy- and Foot Ulcer-Specific Quality of Life instrument (Neuro QOL) is used worldwide to assess the QOL of diabetic patients with peripheral neuropathy. There is no Arabic version of NeuroQOL for use in Egypt.

The study design will be a cross-cultural validation of Neuro Qol the Arabic version for patients with DFUs. Three expert panels were involved in this study to test the face and content validity of Neuro Qol Arabic version. All experts had experience of not less than 10 years or at least a master's degree in physical therapy; a major part of their work is with Arabic population; and they were also fluent in Arabic and English.

Ten patients per item were chosen to estimate the sample size for testing the psychometric properties of the Neuro Qol Arabic version. So 290 patients (145 male patients and 145 female patients), were chosen according to the following criteria: Their age ranged between 18-70 years , with type 2 diabetes referred by physician, conscious and ambulant, and being able to read and write in Arabic.

Patients suffering from congenital deformities, fixed spinal deformity, rheumatoid arthritis, bone disease, or infection were excluded from the study.

Participants will be identified, approached, and recruited from outpatient clinics at the Faculty of Physical Therapy, Nahda University, and El-Salam University. The study will be advertised through posters and word of mouth. Participants will receive a participant information sheet and a self-screening eligibility form, and they will be asked to contact the Principal Investigator (SG) no sooner than 48 hours if they wish to volunteer to participate in the study, which consisted of two visits to the clinic.

During study visit 1, participants will be briefed about the study, screened for eligibility, and enrolled in the study by signing a consent form.

Demographic data, such as age, weight, and height, will also be collected to describe the sample. The principal investigator will apply the clinical examination for the foot and assess any problems such as lost or reduced feeling in your extremities, pain, discomfort, and/or ulcers (open sores) on your feet, and, in some cases, unsteadiness while walking or standing. Participants will then complete the Arabic NeuroQOL. A nurse assisted participants with reading difficulties.

Participants will return for study visit 2 after 7-14 days and will complete the Michigan Diabetic Neuropathy Scale (MDNS)-Arabic version. Participants will also be required to report other symptoms and complications associated with diabetes.

The translation process will follow the Principles of Good Practice for the Translation and Cultural Adaptation Process for Patient-Reported Outcome Measures using the following steps:

1. Preparation: Four bilingual translators who are fluent in Arabic and English will be selected. Three translators are clinicians and one translator is a university academic.
2. Forward translation: the NeuroQOL will be given to all translators to translate into Arabic.
3. Reconciliation: The four translated documents will be shared between all translators, and discrepancies, ambiguities, and issues arising will be discussed and resolved and a final draft Arabic version of the NeuroQOL will be produced.
4. Backward translation and review: The final draft Arabic version of the NeuroQOL will be translated back into English by a translator who had not been involved in forward translation and who was blind to the original English version of the NeuroQOL.
5. Harmonization, cognitive debriefing and reviewing of results: The back-translated The English version of the NeuroQOL will be compared with the original NeuroQOL, and discrepancies, ambiguities, and typographic and/or grammatical errors will be discussed within the group and in the final draft of the Arabic version.
6. Proofreading and final report: When the authenticity of the translation has been agreed upon by consensus, the final version of the Arabic-NeuroQOL will be produced.

ELIGIBILITY:
Inclusion Criteria:

* Arabic is their first language The absence of any other neurological diagnosis affecting the sensory and motor system, such as stroke or multiple sclerosis
* Age ranges between 18 and 70 years,
* History of DM diagnosed by a physician and confirmed by either hemoglobin A1c ≥6.5% or the use of hypoglycemic agents.

Exclusion Criteria:

* A hospital inpatient
* Had pre-existing comorbidities such as cancer, shingles or other neuropathic pain entity that predated diabetes or can mimic or cause a neuropathic pain that is not arising as a result of diabetes.
* Pregnant patients as diabetes may be of gestational type
* Had recently experienced physical trauma that may have contributed to neuropathic pain had trauma or dermatological diseases of the skin as this could affect skin sensitivity (e.g. wounds, psoriasis and eczema).

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study design will be a cross-cultural validation of Neuro Qol the Arabic version for patients with DFUs.
  Participants will be identified, approached, and recruited from outpatient clinic at Faculty of Physical Therapy, Nahda University and Elsalam university. Ten patients per item were chosen to estimate the sample size for testing the psychometric properties of the Neuro Qol Arabic version (Sousa & Rojjanasrirat, 2011). So 290 patients (145 male patients and 145 female patients), were chosen according to specific criterea.
Sampling Method: Probability Sample
Enrollment: 290 (Estimated)
Dates: Start 2025-02-13 (Actual); Primary Completion 2025-12-20 (Estimated); Study Completion 2026-01-25 (Estimated)

PRIMARY OUTCOMES:
Cross-cultural validation of the Arabic-translated NEURQOL Questionnaire. | Baseline and through study completion, an average of 6 months.
  Cross-cultural validation involves three main phases: 1) translation and verification of its equivalence; traditional translation simply involves translation of the original instrument by a bilingual researcher or professional translator. 2) empirical verification of the validity of the translated version; it involves the participation of a number of bilingual people familiar with the field in which the instrument is to be used, which also limits the biases of a single researcher. and 3) adaptation of the scores to the cultural context, and the development of standards. It involves having a preliminary translated version of the instrument translated back into the original language by a second person. The discrepancies between the original version and the retranslated version help identify problematic items.
Reliability of the Arabic-translated NEURQOL Questionnaire. | Baseline and through study completion, an average of 6 months.
  It considers the extent to which the questions used in the NeurQoL questionnaire consistently elicit the same results each time it is asked in the same situation on repeated occasions. test-retest reliability. This involves administering the questionnaire to the eligible participants and repeating the survey with the same group at the end of the questionnaire validation. We then compare the responses at the two time points.
Cross-cultural adaptation of the Arabic-translated NEURQOL Questionnaire. | Baseline and through study completion, an average of 6 months.
  The process of translating and adapting questionnaires from one cultural context to another involves much more than converting the items from the source language to the target language. The questionnaire must be equivalent to the original, considering the new cultural context in which it will be applied. After translation, the scales were evaluated in meetings of a committee of experts in different scientific fields of interest, translators, and language professors. The updated questionnaire was then sent to six experts to assess the relevance of each item, the language, and the adopted response scales, and then to participants from the academic community and organizations human resources to improve item clarity.

CONTACTS AND LOCATIONS:
Overall Officials: Engy BadrEldin S Moustafa, PhD, Principal Investigator — Faculty of Physical Therapy, Cairo University, Egypt
Locations (1):
- Faculty of Physical Therapy, Cairo University, Cairo, Giza Governorate, Egypt